CLINICAL TRIAL: NCT01896336
Title: National Study, Phase IV, Single-center, Double-blind, Randomized, Parallel, Controlled by 10 mg Oral Zolpidem, in Evaluating the Efficacy and Safety of Zolpidem 5 mg Sublingual in the Induction and Maintenance of Sleep in Patients With Primary Insomnia
Brief Title: Efficacy and Safety of 5 mg Sublingual Zolpidem vs 10mg Oral Zolpidem in the Induction and Maintenance of Sleep in Patients With Primary Insomnia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: EMS (Industry)
Collaborators: Associação Fundo de Incentivo à Pesquisa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZPDEMS1011
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Primary Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5mg sublingual Zolpidem hemitartrate (Experimental): 1 QD
  Interventions: Drug: Zolpidem Hemitartrate
- 10 mg oral Zolpidem hemitartrate (Active Comparator): 1 QD.
  Interventions: Drug: Zolpidem Hemitartrate

INTERVENTIONS:
Drug: Zolpidem Hemitartrate — Patz - 5mg sublingual zolpidem hemitartrate
  1 QD
  Stilnox - 10mg oral zolpidem hemitartrate
  1 QD
  Other Names: Patz - 5mg sublingual zolpidem hemitartrate; Stilnox - 10mg oral zolpidem hemitartrate

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of sublingual zolpidem presentation 5 mg in the induction of sleep in patients with primary insomnia.

DETAILED DESCRIPTION:
* National study, phase IV, single-center, double-blind, randomized, parallel, controlled by zolpidem 10mg oral.
* Experiment duration: 93 days.
* 05 visits (days -3, 0, 15, 45 and 90).
* Efficacy will be evaluated for: Sleep induction and the maintenance of sleep.
* Adverse events evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women aged between 20 and 64 years;
* Diagnosis of primary insomnia according to criteria defined by DSM-IV;
* Difficulty in maintaining sleep and waking up until 3 am;
* Not having used any psychoactive drug in the last 30 days prior to their inclusion in the study;
* Signature of IC.

Exclusion Criteria:

* Previous history of serious medical illness, neurological or psychiatric disorder;
* Allergy or hypersensitivity to zolpidem;
* Obstructive Sleep Apnea syndrome;
* Polysomnography with apnea and hypopnea index >10/hour or PLM >15/h;
* Other secondary sleep disorders;
* History of substance abuse or dependence;
* History of daily consumption of alcoholic beverages;
* Pregnancy, lactation or refusal to use safe contraceptive methods during the study.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2013-02-18 (Actual); Primary Completion 2013-11-11 (Actual); Study Completion 2013-12-10 (Actual)

PRIMARY OUTCOMES:
Efficacy will be measured by sleep induction and maintenance. | 90 days
  Sleep induction is measured by time to sleep after administration of the investigational product.
  The maintenance will be measured by the use of medication in the middle of the night and also by the elapsed time to sleep after administration of the investigational drug.

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences | 90 days
  Adverse events will be collected and followed in order to evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Dalva R Poyares, MD, Principal Investigator — Associacao Fundo de Incentivo a Psicofarmcologia
Locations (1):
- AFIP, São Paulo, Sâo Paulo, Brazil

REFERENCES:
- [Derived] Castro LS, Otuyama LJ, Fumo-Dos-Santos C, Tufik S, Poyares D. Sublingual and oral zolpidem for insomnia disorder: a 3-month randomized trial. Braz J Psychiatry. 2020 Apr;42(2):175-184. doi: 10.1590/1516-4446-2019-0389. Epub 2019 Dec 20. PMID 31859791